CLINICAL TRIAL: NCT06787664
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of BL-B01D1 for Injection in Patients With Locally Advanced or Metastatic Chordoma
Brief Title: A Study of BL-B01D1 in Patients With Locally Advanced or Metastatic Chordoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-209
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Chordoma
MeSH Terms: conditions — Chordoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-B01D1 (Experimental): Participants receive BL-B01D1 in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507

SUMMARY:
This is an open-label, multicenter phase II study to evaluate the safety, efficacy and pharmacokinetic characteristics of BL-B01D1 for Injection in patients with locally advanced or metastatic chordoma.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Gender is not limited;
3. Age: ≥18 years old and ≤75 years old;
4. Locally advanced (unresectable) or metastatic chordoma confirmed by histopathology;
5. ECOG ≤2;
6. The expected survival time as judged by the investigator was ≥3 months;
7. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
8. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
9. Organ function level must meet the requirements;
10. Coagulation function: international normalized ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5ULN;
11. Urine protein ≤2+ or < 1000mg/24h;
12. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before starting treatment, a serum or urine pregnancy test must be negative, and the patient must not be lactating; All enrolled patients should take adequate barrier contraception during the entire treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Chemotherapy, biological therapy, immunotherapy, etc. within 4 weeks or 5 half-lives before the first dose, small molecule targeted therapy within 5 days, and palliative radiotherapy within 2 weeks;
2. A history of central nervous system hemorrhage/infarction requiring treatment within 6 months before enrollment;
3. History of severe heart disease and cerebrovascular disease;
4. QT prolongation, complete left bundle branch block, III degree atrioventricular block, severe arrhythmia;
5. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening; Infusion-related thrombosis was excluded;
6. Active autoimmune and inflammatory diseases;
7. Other malignant tumors that progressed or required treatment within 5 years before the first dose;
8. Poorly controlled hypertension (systolic blood pressure after adequate medical therapy > 150 mmHg or diastolic blood pressure > 100 mmHg);
9. Poor glycemic control;
10. Patients with a previous history of ILD requiring hormone therapy, or current ILD or ≥G2 radiation pneumonitis, or suspected to have such a condition during screening;
11. Complicated with pulmonary diseases leading to clinically severe respiratory function impairment;
12. Patients with a history of allergy to recombinant humanized or human-mouse chimeric antibodies or to any of the excipients of BL-B01D1;
13. Received previous organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
14. Human immunodeficiency virus antibody positive, active tuberculosis, active hepatitis B virus infection or active hepatitis C virus infection;
15. Had a serious infection within 4 weeks before the first dose of study drug; Indications of active pulmonary infection within 2 weeks before the first dose of study drug;
16. Imaging examination indicated that the tumor had invaded or enveloped the large blood vessels of the chest, neck, abdomen, ilium, and pharynx, except that the investigator thought that it would not affect the patient's medication;
17. With a history of psychotropic drug abuse and inability to quit or a history of severe neurological or psychiatric illness;
18. Serious unhealed wound, ulcer, or fracture within 4 weeks before signing the informed consent;
19. Clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
20. Patients scheduled for vaccination or receiving live vaccine within 28 days before the first dose;
21. Had participated in another clinical trial within 4 weeks before the first dose;
22. Other circumstances that the investigator deemed inappropriate for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-B01D1 to the first date of either disease progression or death, whichever occurs first.
Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of BL-B01D1 will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of BL-B01D1 will be investigated.
Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of BL-B01D1 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Frequency of anti-BL-B01D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China